CLINICAL TRIAL: NCT02873871
Title: Effect of Two Compression Devices on the Occurrence of Artery Occlusion After Transradial Cardiac Catheterization: Randomized Clinical Trial
Brief Title: Comparison of 2 Hemostasis Techniques After Transradial Coronary
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 49237115.5.0000.5327.
Record Dates: First submitted 2016-04-10; First posted 2016-08-22 (Estimated); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Coronary Artery Disease With Myocardial Infarction
MeSH Terms: conditions — Coronary Artery Disease, Autosomal Dominant, 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (Other): Standardized compressive dressing
  Interventions: Device: Standardized compressive dressing
- Intervention group (Experimental): Hemostasis with TerumoBand®
  Interventions: Device: Hemostasis with TerumoBand®

INTERVENTIONS:
Device: Standardized compressive dressing — Standardized compressive dressing
  Arms: Control group
Device: Hemostasis with TerumoBand® — Hemostasis with TerumoBand®
  Arms: Intervention group

SUMMARY:
Randomized clinical trial to compare radial artery patency after transradial coronary catheterization using 2 different hemostasis techniques. Patients submitted to diagnostic or therapeutic coronary catheterization will be prospectively enrolled in this single-center trial and will be randomized to radial hemostasis with TerumoBand® or a standardized compressive dressing with gauze and elastic bandage.

DETAILED DESCRIPTION:
Randomized clinical trial to compare radial artery patency after transradial coronary catheterization using 2 different hemostasis techniques. Patients submitted to diagnostic or therapeutic coronary catheterization will be prospectively enrolled in this single-center trial and will be randomized to radial hemostasis with TerumoBand® or a standardized compressive dressing with gauze and elastic bandage.

Interventions: Radial hemostasis with TerumoBand® and Radial hemostasis with a standardized compressive dressing

ELIGIBILITY:
Inclusion Criteria:

* Adult patients submitted to elective or urgent coronary catheterization who presented with a A, B or C curve on oximetry test before the procedure

Exclusion Criteria:

* Inability to understand the study and sign the informed consent form

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Radial artery occlusion evaluated using Barbeau's test | up to 3 hours
  test immediately after hemostasis compression device withdrawal

SECONDARY OUTCOMES:
Vascular complications | up to 3 hours
  Clinical assesment
Radial access site pain | up to 3 hours
  standardized scale

CONTACTS AND LOCATIONS:
Overall Officials: Eneida Rejane Rabelo da Silva, RN, MSc, ScD, Study Chair — Hospital de Clinicas de Porto Alegre
Locations (1):
- Universidade Federal do Rio Grande do Sul - Post Graduated Program, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided